CLINICAL TRIAL: NCT05262452
Title: Therapeutic Efficacy and Safety of Concurrent FOLFIRINOX Plus HIFU for Locally Advanced/Borderline Resectable Pancreatic Cancer: A Prospective Single-center, Single-arm, Investigator-initiated, Open-labeled, Exploratory Clinical Trial
Brief Title: Concurrent FOLFIRINOX Plus High Intensity Focused Ultrasound for Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Focused Ultrasound Foundation (Other); Synex Consulting Ltd (Unknown)
Responsible Party: Principal Investigator, Jae Young Lee, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-154-1135
Record Dates: First submitted 2021-10-02; First posted 2022-03-02 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer Non-resectable; Chemotherapy Effect; Ultrasound Therapy
Keywords: High-Intensity Focused Ultrasound Therapy,; Combined Modality Therapy; Clinical Trial; Neoadjuvant Therapy; Survival Analysis; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with locally advanced/borderline resectable pancreatic cancer through biopsy and CT/MRI imaging and planned to undergo anti-cancer treatment using FOLFIRINOX
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CureHIFUPanc (Experimental): Patients diagnosed with locally advanced/borderline resectable pancreatic cancer through biopsy and CT/MRI imaging and planned to undergo anti-cancer treatment using FOLFIRINOX
  Interventions: Device: ALPIUS 900, an ultrasound-guided high intensity focused ultrasound system; Drug: FOLFIRINOX regimen

INTERVENTIONS:
Device: ALPIUS 900, an ultrasound-guided high intensity focused ultrasound system — Device to deliver mechanical stress and force to enhance drug delivery, using focused ultrasound
Drug: FOLFIRINOX regimen — a chemotherapy regimen for treatment of advanced pancreatic cancer
  * FOL : folinic acid (leucovorin), a vitamin B derivative that enhances the effects of 5-FU
  * F : 5-FU, a pyrimidine analog and antimetabolite which incorporates into the DNA molecule and stops DNA synthesis
  * IRIN : irinotecan (eloxatin), a platinum-based antineoplastic agent, which inhibits DNA repair and/or DNA synthesis.
  * OX - oxaliplatin (Eloxatin), a platinum-based antineoplastic agent, which inhibits DNA repair and/or DNA synthesis

SUMMARY:
In patients diagnosed with locally advanced pancreatic cancer (LAPC)/borderline resectable pancreatic cancer (BRPC) and planned chemotherapy using FOLFIRINOX, high intensity focused ultrasound (HIFU)/FOLFIRINOX combined treatment is performed on patients who agree to this study. The combined treatment group is treated in parallel with FOLFIRINOX and HIFU for the first four cycles and then CT is taken for reaction evaluation immediately, 2 months, and 4 months after the four-cycle treatment. For the response assessment, the response rate using RECIST ver. 1.1 and operable rate are evaluated and compared with the results of already established FOLFIRINOX single treatment in the investigators' institute. Time-to-progress and overall survival are calculated.

DETAILED DESCRIPTION:
Patients diagnosed with pancreatic cancer through biopsy and diagnosed with LAPC/BRPC through computed tomography (CT) or magnetic resonance imaging (MRI) are referred to this clinical trial. When the referred patients are voluntarily signed a written consent form after hearing sufficient explanations related to this study, the referred patients will be registered for this clinical trial if all criteria for selection/exception are met.

A management log will be prepared for all subjects who have signed a clinical trial agreement and are registered in the study. These management logs are used to assign sequential subject numbers to subjects registered in clinical trials, and subject numbers are assigned 'screening numbers' and 'registration numbers'.

The subjects will visit on the scheduled date to receive chemotherapy and HIFU combined therapy and will be treated in accordance with the following treatment procedures and protocols.

<Visit 1 to Visit 4: Combined Treatment, Cycle 1, Cycle 2, Cycle 3, Cycle 4 ± 14 Days>

The subjects will receive combined treatments with anticancer drugs (FOLFIRINOX) and HIFU (ALPIUS 900) over four cycles over eight weeks. Afterwards, CT for reaction evaluation is taken immediately after 4 cycles (i.e., 2 months after the onset of combined treatment). CT is taken at intervals of two months up to 6 months after the onset of combined treatment.

At the end of each combined treatment, the patient will be observed about adverse events including anticancer drug adverse events and skin change and can be back home or hospitalized for one to two days after collecting blood for blood tests according to doctor's opinion.

<Schedule and procedures for combined treatment>

Perform a total of four treatments every two weeks for eight weeks.

Combined treatment procedure

Subjects are hospitalized and given anti-cancer drugs for about 50 hours in accordance with the standard protocol for anti-cancer treatment. If the medication is canceled or postponed due to the condition of the subject, the HIFU procedure will be canceled or postponed.

After the start of chemotherapy, receive HIFU treatment within 48 hours (30 minutes to 1 hour) and go up to the inpatient ward to monitor for 1 to 2 hours. If adverse events caused by anticancer drugs have not been recovered within 24 hours of administration or adverse events have not been fully recovered from previous HIFU procedures, the HIFU procedure may be canceled or postponed under the judgment of the investigator.

When combined treatment (anti-cancer drug administration) is completed, the subject shall be hospitalized for one to two days or return home depending on the physical condition of the subject.

<Treatment protocol>

Anti-cancer drug administration (FOLFIRINOX one time regimen) Oxaliplatin 85 mg/m2 (Intravenous, IV) Irinotecan 180 mg/m2 (Intravenous, IV) Leucovorin(Folic acid) 400 mg/m2 (Intravenous, IV) 5-fluorouracil 400 mg/m2 (IV push) 5-fluorouracil 2400 mg/m2 (Intravenous, IV) It is administered at the following schedule every two weeks. Day 1 : Oxaliplatin, Irinotecan, Leucovorin, 5-FU (IV-push), 5-FU (IV infusion) Day 2-3 : 5-FU (IV infusion)

The administration of anticancer drugs (FOLFIRINOX therapy) is applied equally to each treatment group and according to the institution's standard procedure. The FOLFIRINOX dose and administration cycle (interval) can be adjusted by the researcher's judgment depending on the condition and progress of the subject. Anti-cancer drugs used in clinical trials are licensed medicines and are used within the scope of permission.

<HIFU treatment (one-time treatment)>

The HIFU procedure is in accordance with the HIFU parameter, and the details of the pre-procedure, procedure, and post-procedure care of the subjects are in accordance with the manufacturer's ALPIUS 900 User Manual.

HIFU parameter

Acoustic Intensity 2.0 kilowatt (kW)/cm2, Duty cycle 1%, Exposure time 3 sec/point, Pulse repetition frequency (PRF) 10 Hz

Immediately, 2 months, and 4 months after completion of the 4th cycle combined treatment, the subjects visit the hospital to conduct the efficacy and safety assessment. The dose-limiting toxicity (DLT) or adverse device effect (ADE) assessment will be evaluated on each planned visit.

Treatment after the end of combined treatment of HIFU/Anticancer drug Subsequent treatment of patients who have completed HIFU/anti-cancer combined treatment in the first 4 cycles is determined and performed according to findings of CT performed after 4 cycles of combined treatment, overall physical condition of patients, and standard care guidelines. The implementation of surgery, continuation of FOLFIRINOX chemotherapy, conversion to other anticancer drugs, and further radiation therapy can be considered as possible treatments. This assessment is conducted after 8 and 12 cycles of treatment if the treatment continues for FOLFIRINOX chemotherapy, and further treatment policies are determined in accordance with the standard care guidelines. If surgery is performed after 8 or 12 cycles, additional cancer or radiotherapy may be performed after surgery according to surgery and pathological findings, and it is required to be determined in accordance with the standard care guidelines.

ELIGIBILITY:
Inclusion Criteria:

All of the following selection criteria must be met before participants can be registered for this clinical trial.

1. Adults over 19-85
2. Persons with a Karnofsky Performance Scale (KPS) of 70 percent or more;
3. A person diagnosed as a tubular adenocarcinoma through biopsy.
4. A person diagnosed with LAPC/BRPC by computed tomography (CT) or magnetic resonance imaging (MRI)
5. A person willing to voluntarily agree to a clinical trial and comply with the test plan

Exclusion Criteria:

The following exclusion criteria may not be registered in clinical trials.

1. The presence of a cystic lesion within pancreatic cancer to be treated with HIFU or at the pancreas adjacent to the pancreatic cancer.
2. The presence of a wide range of scar or surgical clips observed in the passage through the ultrasonic beam.
3. In case proper ultrasound images for HIFU procedures are not shown
4. A person who cannot lie down in a comfortable position.
5. A person who has difficulty communicating
6. A person who has experience in toxic or hypersensitive reactions to FOLFIRINOX anticancer drugs.
7. A person pregnant or breastfeeding
8. Pancreatic cancer patients who have previously been anti-cancer treatment
9. If severe side effects such as aortic rupture, duodenum perforation, gastrointestinal damage or intestinal necrosis are expected due to HIFU procedures.
10. Other cases where participation in this clinical trial is judged inappropriate by the investigator (specific reasons should be recorded in the case report form)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
2-month Tumor Response | immediately after the completion of the four-cycle combined treatment (each cycle is 14 days)
  Based on CT findings taken immediately after completion of the four-cycle combined treatment (each cycle is 14 days), 2-month tumor response is evaluated with complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) according to the Response Evaluation Criteria In Solid Tumors (RECIST, Ver 1.1)
4-month Tumor Response | 4 months after the start of combined treatment
  Based on CT findings taken obtained 4 months after the start of combined treatment, 4-month tumor response is evaluated with complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) according to the Response Evaluation Criteria In Solid Tumors (RECIST, Ver 1.1)
6-month Tumor Response | 6 months after the start of combined treatment
  Based on CT findings taken obtained 6 months after the start of combined treatment, 6-month tumor response is evaluated with complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) according to the Response Evaluation Criteria In Solid Tumors (RECIST, Ver 1.1)
Percentage of subjects that were subject to surgical resection | 4 months or 6 months after the start of the combined treatment
  When surgery is determined according to American Joint Committee on Cancer (AJCC), 8 edition guidelines based on computed tomography (CT) images taken 4 months or 6 months after the start of the combined treatment, the percentage of subjects who were able to be operated on compared to the total number of registered subjects is calculated.

SECONDARY OUTCOMES:
Time-to-Progression | from the date of diagnosis of pancreatic cancer or from the start date of combined treatment of pancreatic cancer until the date of first documented progression, assessed up to 24 month
  The time taken from the date of diagnosis of pancreatic cancer or from the start date of combined treatment of pancreatic cancer until the date of first documented progression, assessed up to 24 months. Judging by RECIST ver. 1.1
Survival time | from the date of diagnosis of pancreatic cancer or the start date of combined treatment of pancreatic cancer until the date of death from any cause, assessed up to 24 months
  The time taken from the date of diagnosis of pancreatic cancer or the start date of combined treatment of pancreatic cancer until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jae Young Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490
- [Background] Murphy JE, Wo JY, Ryan DP, Jiang W, Yeap BY, Drapek LC, Blaszkowsky LS, Kwak EL, Allen JN, Clark JW, Faris JE, Zhu AX, Goyal L, Lillemoe KD, DeLaney TF, Fernandez-Del Castillo C, Ferrone CR, Hong TS. Total Neoadjuvant Therapy With FOLFIRINOX Followed by Individualized Chemoradiotherapy for Borderline Resectable Pancreatic Adenocarcinoma: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Jul 1;4(7):963-969. doi: 10.1001/jamaoncol.2018.0329. PMID 29800971
- [Background] Choi YH, Lee SH, You MS, Shin BS, Paik WH, Ryu JK, Kim YT, Kwon W, Jang JY, Kim SW. Prognostic Factors for Patients with Borderline Resectable or Locally Advanced Pancreatic Cancer Receiving Neoadjuvant FOLFIRINOX. Gut Liver. 2021 Mar 15;15(2):315-323. doi: 10.5009/gnl19182. PMID 32235008
- [Background] Hackert T, Sachsenmaier M, Hinz U, Schneider L, Michalski CW, Springfeld C, Strobel O, Jager D, Ulrich A, Buchler MW. Locally Advanced Pancreatic Cancer: Neoadjuvant Therapy With Folfirinox Results in Resectability in 60% of the Patients. Ann Surg. 2016 Sep;264(3):457-63. doi: 10.1097/SLA.0000000000001850. PMID 27355262
- [Background] Wu F, Wang ZB, Zhu H, Chen WZ, Zou JZ, Bai J, Li KQ, Jin CB, Xie FL, Su HB. Feasibility of US-guided high-intensity focused ultrasound treatment in patients with advanced pancreatic cancer: initial experience. Radiology. 2005 Sep;236(3):1034-40. doi: 10.1148/radiol.2362041105. Epub 2005 Jul 29. PMID 16055692
- [Background] Vidal-Jove J, Perich E, Del Castillo MA. Ultrasound Guided High Intensity Focused Ultrasound for malignant tumors: The Spanish experience of survival advantage in stage III and IV pancreatic cancer. Ultrason Sonochem. 2015 Nov;27:703-706. doi: 10.1016/j.ultsonch.2015.05.026. Epub 2015 May 27. PMID 26044461
- [Background] Marinova M, Huxold HC, Henseler J, Mucke M, Conrad R, Rolke R, Ahmadzadehfar H, Rauch M, Fimmers R, Luechters G, Cuhls H, Radbruch L, Schild HH, Strunk H. Clinical Effectiveness and Potential Survival Benefit of US-Guided High-Intensity Focused Ultrasound Therapy in Patients with Advanced-Stage Pancreatic Cancer. Ultraschall Med. 2019 Oct;40(5):625-637. doi: 10.1055/a-0591-3386. Epub 2018 Apr 17. PMID 29665583
- [Background] Li T, Wang YN, Khokhlova TD, D'Andrea S, Starr F, Chen H, McCune JS, Risler LJ, Mashadi-Hossein A, Hingorani SR, Chang A, Hwang JH. Pulsed High-Intensity Focused Ultrasound Enhances Delivery of Doxorubicin in a Preclinical Model of Pancreatic Cancer. Cancer Res. 2015 Sep 15;75(18):3738-46. doi: 10.1158/0008-5472.CAN-15-0296. Epub 2015 Jul 27. PMID 26216548
- [Background] Lee ES, Lee JY, Kim H, Choi Y, Park J, Han JK, Choi BI. Pulsed high-intensity focused ultrasound enhances apoptosis of pancreatic cancer xenograft with gemcitabine. Ultrasound Med Biol. 2013 Nov;39(11):1991-2000. doi: 10.1016/j.ultrasmedbio.2013.06.004. Epub 2013 Aug 22. PMID 23972483
- [Background] Lee JY, Choi BI, Ryu JK, Kim YT, Hwang JH, Kim SH, Han JK. Concurrent chemotherapy and pulsed high-intensity focused ultrasound therapy for the treatment of unresectable pancreatic cancer: initial experiences. Korean J Radiol. 2011 Mar-Apr;12(2):176-86. doi: 10.3348/kjr.2011.12.2.176. Epub 2011 Mar 3. PMID 21430934
- [Background] Rapoport N, Payne A, Dillon C, Shea J, Scaife C, Gupta R. Focused ultrasound-mediated drug delivery to pancreatic cancer in a mouse model. J Ther Ultrasound. 2013 Jul 1;1:11. doi: 10.1186/2050-5736-1-11. eCollection 2013. PMID 25516800
- [Background] Park EJ, Ahn YD, Lee JY. In vivo study of enhanced chemotherapy combined with ultrasound image-guided focused ultrasound (USgFUS) treatment for pancreatic cancer in a xenograft mouse model. Eur Radiol. 2018 Sep;28(9):3710-3718. doi: 10.1007/s00330-018-5355-9. Epub 2018 Mar 29. PMID 29600477
- [Background] Yu MH, Lee JY, Kim HR, Kim BR, Park EJ, Kim HS, Han JK, Choi BI. Therapeutic Effects of Microbubbles Added to Combined High-Intensity Focused Ultrasound and Chemotherapy in a Pancreatic Cancer Xenograft Model. Korean J Radiol. 2016 Sep-Oct;17(5):779-88. doi: 10.3348/kjr.2016.17.5.779. Epub 2016 Aug 23. PMID 27587968
- [Background] Kim JH, Kim H, Kim YJ, Lee JY, Han JK, Choi BI. Dynamic contrast-enhanced ultrasonographic (DCE-US) assessment of the early response after combined gemcitabine and HIFU with low-power treatment for the mouse xenograft model of human pancreatic cancer. Eur Radiol. 2014 Sep;24(9):2059-68. doi: 10.1007/s00330-014-3260-4. Epub 2014 Jun 25. PMID 24962825
- [Background] Yoo C, Lee SS, Song KB, Jeong JH, Hyung J, Park DH, Song TJ, Seo DW, Lee SK, Kim MH, Lee SS, Kim JH, Jin HS, Park JH, Hwang DW, Lee JH, Lee W, Chang HM, Kim KP, Ryoo BY, Kim SC. Neoadjuvant modified FOLFIRINOX followed by postoperative gemcitabine in borderline resectable pancreatic adenocarcinoma: a Phase 2 study for clinical and biomarker analysis. Br J Cancer. 2020 Aug;123(3):362-368. doi: 10.1038/s41416-020-0867-x. Epub 2020 May 20. PMID 32433600
- [Background] Janssen QP, Buettner S, Suker M, Beumer BR, Addeo P, Bachellier P, Bahary N, Bekaii-Saab T, Bali MA, Besselink MG, Boone BA, Chau I, Clarke S, Dillhoff M, El-Rayes BF, Frakes JM, Grose D, Hosein PJ, Jamieson NB, Javed AA, Khan K, Kim KP, Kim SC, Kim SS, Ko AH, Lacy J, Margonis GA, McCarter MD, McKay CJ, Mellon EA, Moorcraft SY, Okada KI, Paniccia A, Parikh PJ, Peters NA, Rabl H, Samra J, Tinchon C, van Tienhoven G, van Veldhuisen E, Wang-Gillam A, Weiss MJ, Wilmink JW, Yamaue H, Homs MYV, van Eijck CHJ, Katz MHG, Groot Koerkamp B. Neoadjuvant FOLFIRINOX in Patients With Borderline Resectable Pancreatic Cancer: A Systematic Review and Patient-Level Meta-Analysis. J Natl Cancer Inst. 2019 Aug 1;111(8):782-794. doi: 10.1093/jnci/djz073. PMID 31086963
- [Background] Suker M, Beumer BR, Sadot E, Marthey L, Faris JE, Mellon EA, El-Rayes BF, Wang-Gillam A, Lacy J, Hosein PJ, Moorcraft SY, Conroy T, Hohla F, Allen P, Taieb J, Hong TS, Shridhar R, Chau I, van Eijck CH, Koerkamp BG. FOLFIRINOX for locally advanced pancreatic cancer: a systematic review and patient-level meta-analysis. Lancet Oncol. 2016 Jun;17(6):801-810. doi: 10.1016/S1470-2045(16)00172-8. Epub 2016 May 6. PMID 27160474
- [Background] Rombouts SJ, Walma MS, Vogel JA, van Rijssen LB, Wilmink JW, Mohammad NH, van Santvoort HC, Molenaar IQ, Besselink MG. Systematic Review of Resection Rates and Clinical Outcomes After FOLFIRINOX-Based Treatment in Patients with Locally Advanced Pancreatic Cancer. Ann Surg Oncol. 2016 Dec;23(13):4352-4360. doi: 10.1245/s10434-016-5373-2. Epub 2016 Jul 1. PMID 27370653

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT05262452/Prot_SAP_000.pdf